CLINICAL TRIAL: NCT00191477
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 3 Multicenter Study of Immediate Postoperative Instillation of Gemcitabine in Patients With Superficial Transitional Cell Carcinoma of the Bladder
Brief Title: Instillation of Gemcitabine in Patients With Superficial Bladder Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped early for futility reasons.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6138; B9E-MC-S274
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2009-10-28 (Estimated); Last update posted 2009-10-28 (Estimated); Status verified 2009-09

CONDITIONS: Bladder Neoplasms
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: Gemcitabine
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gemcitabine — 2000 mg, intravesicular instillation x 1 immediately post transurethral resection of the bladder tumor (TUR-BT)
  Other Names: LY 188011; Gemzar
  Arms: A
Drug: Placebo — intravesicular instillation x 1 immediately post transurethral resection of the bladder tumor (TUR-BT)
  Arms: B

SUMMARY:
A randomized, double-blind, placebo-controlled Phase 3 multicenter study to assess the efficacy and safety of intravesical instillation of gemcitabine versus placebo immediately after transurethral resection of the bladder tumor.

ELIGIBILITY:
Inclusion Criteria:

* Clinical evidence of superficial transitional cell carcinoma of the bladder
* Males or females at least 18 years of age
* Karnofsky Performance Status greater than or equal to 70%
* Patient compliance and geographic proximity that allow adequate follow-up
* Female patients with reproductive potential must use a reliable contraceptive method if appropriate (for example, intrauterine device [IUD], birth control pills, or barrier device) during the study. Female patients with reproductive potential must have a negative serum pregnancy test within 7 days of study enrollment.
* Signed informed consent.

Exclusion Criteria:

* Clinical evidence of muscle-invasive or locally advanced bladder cancer
* Clinical evidence of upper urinary tract tumor
* Distant metastases
* Other malignancies within the last 2 years, except non-melanotic skin tumors, carcinoma in situ of the cervix or organ-confined prostate cancer after curative therapy
* Severe concomitant psychiatric disease
* Febrile, active infection
* Other serious concomitant disorders that would compromise the safety of the patient or his/her ability to complete the study according to the protocol, at the discretion of the investigator (for example, unstable angina pectoris, uncontrolled diabetes mellitus)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2004-01; Primary Completion 2008-03 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY(1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5PM Eastern time (UTC/GMT - 5 hours, EST), Study Chair — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559,1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physici, Reinfeld, Germany

REFERENCES:
- [Derived] Han MA, Maisch P, Jung JH, Hwang JE, Narayan V, Cleves A, Hwang EC, Dahm P. Intravesical gemcitabine for non-muscle invasive bladder cancer. Cochrane Database Syst Rev. 2021 Jun 14;6(6):CD009294. doi: 10.1002/14651858.CD009294.pub3. PMID 34125951
- [Derived] Bohle A, Leyh H, Frei C, Kuhn M, Tschada R, Pottek T, Wagner W, Knispel HH, von Pokrzywnitzki W, Zorlu F, Helsberg K, Lubben B, Soldatenkova V, Stoffregen C, Buttner H; S274 Study Group. Single postoperative instillation of gemcitabine in patients with non-muscle-invasive transitional cell carcinoma of the bladder: a randomised, double-blind, placebo-controlled phase III multicentre study. Eur Urol. 2009 Sep;56(3):495-503. doi: 10.1016/j.eururo.2009.06.010. Epub 2009 Jun 21. PMID 19560257
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 355 participants were enrolled and randomized (included here in disposition); however, due to study design, only 328 (N=166 Gemcitabine and N=162 Placebo) actually received study drug (Full Analysis Set).
Period: Overall Study
Arm/Group | Gemcitabine | Placebo
Started | 179 | 176
Received Study Drug | 166 | 162
Completed | 41 | 47
Not Completed | 138 | 129
Not completed — Tumor Recurrence | 49 | 48
Not completed — Death, Study Disease | 1 | 1
Not completed — Death, Other Cause | 3 | 6
Not completed — Lost to Follow-up | 23 | 21
Not completed — Protocol Violation | 1 | 1
Not completed — Treatment Change | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Other | 2 | 0
Not completed — Not Eligible | 41 | 38
Not completed — Pathological Specimen Lost | 1 | 0
Not completed — Discontinued Prior to Instillation | 13 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gemcitabine | Placebo | Total
Number analyzed (Participants) | 166 | 162 | 328
Age Continuous [Mean (Standard Deviation); unit: years] | 63.2 (11.9) | 66.3 (11.0) | 64.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 26 | 65.0
  Male | 127 | 136 | 263.0
Region of Enrollment [Number; unit: participants]
  Germany | 131 | 126 | 257.0
  Turkey | 35 | 36 | 71.0
Karnofsky Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Rating occurs in steps of 10 score points (0=death, 10, 20,....up to 100=Normal no complaints, no evidence of disease). Lower scores indicate poorer patient condition.
  participants
    70 - Unable to carry on normal activity | 1 | 1 | 2.0
    80 - Activity with effort; some signs of disease | 13 | 7 | 20.0
    90 - Normal activity; minor signs of disease | 33 | 49 | 82.0
    100 - Normal no complaints; no evidence of disease | 118 | 104 | 222.0
    Unspecified | 1 | 1 | 2.0
Newly Diagnosed versus Recurrent Disease [Number; unit: participants]
  Recurrent Disease | 43 | 40 | 83.0
  Newly Diagnosed | 123 | 122 | 245.0
Race/Ethnicity [Number; unit: participants]
  White | 166 | 162 | 328
Results of Initial Transurethral Resection of a Bladder Tumor (TUR-BT): Number of Visible Lesions [Number; unit: participants] — The initial TUR-BT was the first and mandatory TUR-BT during the study. An optional second TUR-BT was allowed.
  participants
    No Lesions (No Specific Sites Documented) | 4 | 5 | 9.0
    1 Lesion | 87 | 96 | 183.0
    2 Lesions | 42 | 27 | 69.0
    3 Lesions | 18 | 14 | 32.0
    4 Lesions | 7 | 10 | 17.0
    >=5 Lesions | 8 | 10 | 18.0
Results of Transurethral Resection of Bladder Tumor (TUR-BT): Final Pathological Disease Stage [Number; unit: participants] — Worst staging of the initial and optional second transurethral resection of bladder tumor.
  participants
    pTx: Primary Tumor Cannot be Assessed | 3 | 0 | 3.0
    pT0: No Evidence of Primary Tumor | 0 | 0 | 0.0
    pTa: Noninvasive Papillary Carcinoma | 93 | 88 | 181.0
    pT1: Tumor Invades Subepithelial Connective Tissue | 31 | 36 | 67.0
    >=pT2: Tumor Invades Wider Area | 12 | 10 | 22.0
    Cis: Carcinoma in situ ("Flat Tumor") | 5 | 6 | 11.0
    No Malignancy | 21 | 22 | 43.0
    Unspecified | 1 | 0 | 1.0
Results of Transurethral Resection on a Bladder Tumor (TUR-BT): Final Disease Grade [Number; unit: participants] — Worst grading of the initial and optional second transurethral resection of bladder tumor.
  participants
    G1 - Well Differentiated | 59 | 66 | 125.0
    G2 - Moderately Differentiated | 50 | 48 | 98.0
    G3 - Poorly Differentiated | 25 | 24 | 49.0
    G4 - Undifferentiated | 3 | 1 | 4.0
    GX - Unknown | 8 | 1 | 9.0
    Unspecified | 21 | 22 | 43.0

OUTCOME MEASURES:

1. Primary Outcome: Recurrence-Free Survival (RFS)
Description: Defined as the time from study enrollment to the date of the first procedure confirming histopathological recurrence or disease progression or death from any cause. Recurrence-free survival (RFS) was censored at the date of the last follow-up visit for participants who were still alive and who had no recurrence/progression.
Time Frame: Surgery to recurrence or death (Follow-up assessments were performed at 3 and 6 months after the first TUR-BT, and every 6 months thereafter, until recurrence/progression of disease, or until the end of study, up to 24 months)
Population: This is the Full Analysis Set population and contains all randomized participants who received the single instillation of Gemcitabine or Placebo.
Measure: Median (Full Range); unit: Months
Arm/Group | Gemcitabine | Placebo
Number analyzed (Participants) | 166 | 162
Months | 37.2 [0.0 to 45.9] | 40.2 [0.0 to 42.2]
Statistical Analysis 1: Comparison: Gemcitabine vs Placebo; Sample-size calculation based on estimated 1-year recurrence-free survival (RFS) rates of 63% (gemcitabine) and 50% (placebo). 191 critical events were required to detect a difference in RFS (80% power, log-rank test, alpha=0.050). Sample size of 328 patients with clinical evidence of superficial bladder cancer needed to observe these 191 events within a 24-month follow-up period, assuming 246 of these patients would receive instillation and have histopathological diagnosis of pTa/pT1(G1-3/Gx); Test type: Superiority or Other; p = 0.777, Log Rank — Only 87 recurrences and 7 deaths were documented at planned end of follow-up. The study was stopped early for futility reasons based on an interim analysis using pre-defined stopping boundaries for the hazard ratio (HR) of RFS; Hazard Ratio (HR) = 0.946, 95% CI [0.643 to 1.392]

2. Post Hoc Outcome: Percentage of Participants Without Tumor Recurrence
Description: Because median time to recurrence was not reached, percentage of participants without event was estimated using Kaplan-Meier method. Time to recurrence was censored on date of death for patients who died, and on date of last visit for patients who were alive, without recurrence.
Time Frame: Surgery to recurrence (Follow-up assessments were performed at 3 and 6 months after the first TUR-BT, and every 6 months thereafter, until recurrence/progression of disease, or until the end of study, up to 24 months)
Population: Efficacy Eligible population contains the Full Analysis Set participants with histopathologically confirmed papillary superficial transitional cell carcinoma of the bladder.
Measure: Number; unit: percentage of participants
Arm/Group | Gemcitabine | Placebo
Number analyzed (Participants) | 124 | 124
percentage of participants
  Recurrence-Free at 12 Months | 78.4 [56.4 to 74.5] | 76.9 [53.9 to 71.9]
  Recurrence-Free at 24 Months | 66.3 | 63.7

3. Post Hoc Outcome: Percentage of Participants in Subgroups With Recurrence-Free Survival (RFS) at 12 and 24 Months
Description: RFS rate was estimated using Kaplan-Meier method. RFS was analyzed in different subgroups based on risk, disease status, and concomitant Bacillus Calmette-Guerin (BCG) instillations. Risk: Grading (G1,G2,G3) was performed according to American Joint Committee on Cancer Staging Criteria for Bladder Cancer. Newly diagnosed disease: Initial diagnosis at study entry. Recurrent disease: history of at least one superficial bladder tumor that was surgically treated and relapsed prior to study entry. With BCG: received at least one instillation of BCG during study. Without BCG: didn't receive BCG.
Time Frame: as for outcome 1
Population: Efficacy Eligible population consists of the Full Analysis Set (randomized) participants with histopathologically confirmed papillary superficial transitional cell carcinoma of the bladder.
Measure: Number; unit: percentage of participants
Arm/Group | Gemcitabine | Placebo
Number analyzed (Participants) | 124 | 124
percentage of participants
  Low Risk (G1/G2) - 12 Months (N=106, N=109) | 78.5 [68.9 to 85.4] | 78.4 [69.1 to 85.2]
  Low Risk (G1/G2) - 24 Months (N=106, N=109) | 63.9 | 64.3
  High Risk (G3) - 12 Months (N=13, N=14) | 66.7 [33.7 to 86.0] | 42.4 [13.7 to 69.1]
  High Risk (G3) - 24 Months (N=13, N=14) | 57.1 | 31.8
  Newly Diagnosed Disease - 12 Months (N=94, N=98) | 79.3 [69.1 to 86.4] | 79.8 [69.9 to 86.8]
  Newly Diagnosed Disease - 24 Months (N=94, N=98) | 65.4 | 63.6
  Recurrent Disease - 12 Months (N=30, N=26) | 72.2 [50.4 to 85.7] | 58.9 [37.1 to 75.5]
  Recurrent Disease - 24 Months (N=30, N=26) | 59.5 | 50.5
  With BCG - 12 Months (N=13, N=21) | 61.5 [30.8 to 81.8] | 79.4 [54.0 to 91.7]
  With BCG - 24 Months (N=13, N=21) | 49.2 | 63.5
  Without BCG - 12 Months (N=111, N=103) | 79.9 [70.6 to 86.6] | 74.5 [64.4 to 82.1]
  Without BCG - 24 Months (N=111, N=103) | 65.8 | 60.1

4. Secondary Outcome: Time to Recurrence
Description: Time from enrollment to first confirmation of histopathological recurrence or disease progression. Time to recurrence was censored on date of death for patients who died, and on date of last visit for patients who were alive, without recurrence.
Time Frame: as for outcome 2
Population: Because median time to recurrence was not reached in placebo arm, percentages of participants without recurrence are reported as post-hoc outcome measure (see #5. Post-hoc Outcome Measure). Efficacy Eligible population consists of randomized patients with histopathologically confirmed papillary superficial transitional cell carcinoma of bladder.
Measure: Median (Full Range); unit: months
Arm/Group | Gemcitabine | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Recurrence-Free Survival (RFS) in Subgroups
Description: Defined as the time from study enrollment to the date of the first procedure confirming histopathological recurrence or disease progression or death from any cause. Recurrence-free survival was censored at the date of the last follow-up visit for participants who were still alive and who had no recurrence/progression.
Time Frame: as for outcome 1
Population: Because median time for RFS was not reached in all subgroups, patients (%) with RFS are reported as post-hoc outcome #6. There was no statistically significant difference between treatment arms in any subgroup. Population consists of randomized patients with histopathologically confirmed papillary superficial transitional cell carcinoma of bladder.
Measure: Median (Full Range); unit: months
Arm/Group | Gemcitabine | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Tumor Recurrence Type
Description: Tumor recurrence type (superficial, stage pTA or pT1; or muscle-invasive, stage≥pT2) was classified according to American Joint Committee on Cancer Staging Criteria for Bladder Cancer (AJCC Cancer Staging Manual, 6th edition).
Time Frame: as for outcome 2
Population: Efficacy Eligible population consists of the Full Analysis Set participants with histopathologically confirmed papillary superficial transitional cell carcinoma of the bladder.
Measure: Number; unit: participants
Arm/Group | Gemcitabine | Placebo
Number analyzed (Participants) | 124 | 124
participants
  No Tumor Recurrence | 76 | 78
  Superficial Tumor - Stage pTa or pT1 | 44 | 45
  Muscle-Invasive Tumor - Any Stage ≥pT2 | 3 | 1
  pTx - Tumor Cannot be Assessed | 1 | 0

ADVERSE EVENTS:
Groups:
- Gemcitabine: Gemcitabine: 2000 mg, intravesicular instillation x 1 immediately post transurethral resection of bladder tumor (TUR-BT)
- Placebo: Placebo: intravesicular instillation x 1 immediately post transurethral resection of bladder tumor (TUR-BT)
Arm/Group | Gemcitabine | Placebo
Serious Adverse Events (participants affected / at risk) | 17/166 | 10/162
Other Adverse Events (participants affected / at risk) | 38/166 | 36/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine (N=166) | Placebo (N=162)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cystoprostatectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Urinary bladder excision (Surgical and medical procedures) | 8 (8) | 5 (5)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine (N=166) | Placebo (N=162)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Double ureter (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Kidney duplex (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 1 (1)
Face oedema (General disorders) | 1 (1) | 0 (0)
Hyperpyrexia (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 5 (5)
Pyrexia (General disorders) | 3 (3) | 1 (1)
Cystitis (Infections and infestations) | 2 (2) | 5 (5)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Urethritis (Infections and infestations) | 2 (2) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Post procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural vomiting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anticholinergic syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (2)
Sleep disorder (Psychiatric disorders) | 1 (1) | 3 (3)
Bladder diverticulum (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder pain (Renal and urinary disorders) | 5 (6) | 3 (4)
Bladder spasm (Renal and urinary disorders) | 1 (1) | 4 (4)
Dysuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral meatus stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral stricture (Renal and urinary disorders) | 0 (0) | 1 (1)
Urge incontinence (Renal and urinary disorders) | 1 (1) | 1 (1)
Vesical tenesmus (Renal and urinary disorders) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Alopecia areata (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urinary bladder excision (Surgical and medical procedures) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was stopped early for futility reasons. In addition, due to limitations in this databank, some original outcome measures are not disclosed. Time to Recurrence and Recurrence-Free Survival in Subgroups had data that were un-estimated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days